CLINICAL TRIAL: NCT04274803
Title: Dose Intralipid Infusion Reduces Pregnancy Complications Caused by Antiphospholipid Antibody Syndrome?
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: no patient enrolled
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ayman S Dawood, MD, Lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INTRALIPID-APS
Record Dates: First submitted 2020-02-15; First posted 2020-02-18 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Antiphospholipid Syndrome in Pregnancy
MeSH Terms: interventions — soybean oil, phospholipid emulsion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intralipid group (Experimental): the patients will receive the conventional basic treatment of APS (Dual low dose aspirin (LDA) (Ezacard 75mg) once daily and Low molecular weight heparin (LMWH) (clexane 4000 IU) injection once daily. In addition intralipid 20% (Frezenius, Clayton, NC, USA) in a dose of 4 ml diluted in 250 ml 0.9% regular saline to be infused IV and to be repeated every 2 weeks all over the pregnancy.
  Interventions: Drug: Intralipid, 20% Intravenous Emulsion
- Standard care group (Active Comparator): the patients will receive the conventional basic treatment of APS (Dual low dose aspirin (LDA) (Ezacard 75mg) once daily and Low molecular weight heparin (LMWH) (clexane 4000 IU) injection once daily.
  Interventions: Drug: Conventional therapy of antiphospholipis syndrome

INTERVENTIONS:
Drug: Intralipid, 20% Intravenous Emulsion — intralipid 20% (Frezenius, Clayton, NC, USA) in a dose of 4 ml diluted in 250 ml 0.9% regular saline to be infused IV and to be repeated every 2 weeks all over the pregnancy.
  Arms: Intralipid group
Drug: Conventional therapy of antiphospholipis syndrome — the conventional basic treatment of APS (Dual low dose aspirin (LDA) (Ezacard 75mg) once daily and Low molecular weight heparin (LMWH) (clexane 4000 IU) injection once daily.
  Arms: Standard care group

SUMMARY:
This study will address the value of adding intralipid infusion in reducing pregnancy complications related to antiphospholipid syndrome

DETAILED DESCRIPTION:
This study will be conducted in the Department of Obstetrics and Gynecology, Tanta University on patients attending the antenatal care clinic and also on patients attending the researchers private clinics for antenatal care. The number of patients enrolled in the study will be 105 patients after application of inclusion and exclusion criteria.

All women wil be thoroughly informed about the study aims and through discussion about the procedure, associated benefits and risks and will sign a written consent.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at booking date who were already diagnosed to have antiphospholipid syndrome (APS) .

Exclusion Criteria:

* Patients with gestational age ≥ 9 weeks
* patients with diagnosed other auto-immune disorder
* patients with chronic hypertension, diabetes mellitus, thyroid disorders,
* patient with renal diseases
* patients who requested to withdraw from the study at any point .

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Fetal loss | within 9 months
  Fetal demise
Premature delivery | Before 37 weeks
  occurrence of preterm labour before 37 weeks
Preeclampsia | > 20 weeks
  Hypertesion, proteiuria and or edema
fetal growth restriction | within 9 months
  Fetal poderal index less than normal

CONTACTS AND LOCATIONS:
Locations (1):
- Adel Elgergawy, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
when approved by ethical committee
Supporting Information: Study Protocol
Time Frame: 9 months